CLINICAL TRIAL: NCT01786889
Title: Identification, Molecular Epidemiology Angiosarcoma of the Liver France
Acronym: ANGIHE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut de Veille Sanitaire (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANGI HE-1110; 2012-A00739-34 (IDRCB Number) (Other: AFSSAPS)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma | interventions — Blood Specimen Collection; Urination; Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with angiosarcoma of the liver (Experimental): Blood and urine collections, questionnaire and telephone interview
  Interventions: Biological: blood and urine; Behavioral: Questionnaire; Behavioral: Telephone interview

INTERVENTIONS:
Biological: blood and urine — Blood collection and urine collection after consent of the patient
Behavioral: Questionnaire — The patient complete the questionnaire alone at home
Behavioral: Telephone interview — The patient will be contacted by the CRA for a telephone interview of around one hour

SUMMARY:
The purpose of this study is to test the feasibility of identifying incident cases of angiosarcoma of the liver from the network NetSarc.

DETAILED DESCRIPTION:
The study involves a questionnaire and a one-hour telephone interview.

Consultation:

* Study proposal
* Information and collection of the patient's and/or parent's written consents
* Blood collection (10ml) and urine collection of the patient and parents if applicable
* Delivery of a specific questionnaire and a stamped envelope (with the address of the coordinator's center). If it's about a child patient or an adolescent under 18 years, 3 questionnaires will be given (1 for each parent and 1 for the child).

At home: Filling the questionnaire by the patient and/or the parents, alone at home and return to the coordinator via the given envelope.

During the study: Collect of the initial biopsies used for the hepatic angiosarcoma's diagnostic.

End of the study: Telephone interview CRA/Patient and/or parents to complete the questionnaires (around one hour). From this data will be reconstitute the residential process of the patient and parents if it's about a child or an adolescent (collection of the successive addresses).

Finally, water collections, according to a defined sampling protocol, at the tap of the different homes and places visited by the patients will be organized by the InvS in relation to the ARS within the scope of water quality controls, in order to evaluate the exposition to vinyl chloride monomer (VCM) by hydric ways.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with angiosarcoma of the liver (angiosarcoma immediately multifocal allowed) diagnosed by histology from the start of the study
* The patient's written Consent

No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06; Primary Completion 2016-09 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of identifying incident cases of angiosarcoma liver from the network NetSarc | At month 36
  Feasibility of identifying incident cases of angiosarcoma of the liver (ASF) from the network NetSarc: number of sheets indicated and returned to the Promoter. 30 cases are expected, the cumulative number of incident cases will be measured over a period of 36 months

SECONDARY OUTCOMES:
Prospective surveillance in France | At month 36
Description of occupational risk factors and environmental | At month 36
  Data will be collected using a questionnaire with:
  * Exhaustive search of all occupational and environmental exposures as known or suspected risk factors for ASF
  * Reconstruction of residential history and haunts each case by means of a collection of successive addresses
Identification of biomarkers associated with human exposure Environmental old and new to vinyl chloride monomer | At 36 month
  Research suggestive of carcinogenesis related to CVM (identified in animal models and cohorts of workers exposed) biomarkers will be made by biological testing (blood and urine) adducts éthénobases kind resulting from the reaction of metabolites with CVM DNA and specific gene mutations k-ras and p53. Exposure to arsenic via the determination of Arsenic urinaire.sera sought.
  The p53 and K-ras genes are also sequences from initial diagnostic biopsies.
Assessment of the amount of vinyl chloride monomèredans successive addresses or nearby for cases without occupational exposure identified | At month 36
  Data will be collected using a questionnaire with:
  - Assessment of the amount of vinyl chloride monomer (VCM) in successive addresses or nearby for cases without occupational exposure identified

CONTACTS AND LOCATIONS:
Overall Officials: LE MOAL Joelle, Dr, Study Director — Institut de Veille Sanitaire_Département Santé Environnement; PENEL Nicolas, MD, Principal Investigator — Centre Oscar Lambret
Locations (12):
- France (12):
  - Institut Bergonié, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la TIMONE, Marseille
  - CRLCC Montpellier, Montpellier
  - Hopital Tenon, Paris
  - Institut de Cancérologie Lucien, Saint-Priest-en-Jarez
  - CHU Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Chu / Hopital Trousseau, Tours

IPD SHARING:
Plan to Share IPD: No